CLINICAL TRIAL: NCT04303377
Title: Early Treatment With evOlocumab in Patients With sT-elevation Myocardial Infarction Undergoing Primary pCi (ExOTIC Study)
Brief Title: Early Treatment With Evolocumab in Patients With ST-elevation Myocardial Infarction
Acronym: ExOTIC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor required early termination of the economic agreement due to a supposed extension of the enrollment period for bureaucracy reasons and for the concomitant Covid -19 Pandemic
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Centro Cardiologico Monzino (Other); Ospedale Bassini Cinisello Balsamo (Unknown); Azienda Ospedaliera Ordine Mauriziano di Torino (Other); Ospedale Policlinico San Martino (Other); Fondazione Poliambulanza Istituto Ospedaliero (Other); Azienda Ospedaliera San Gerardo di Monza (Other); Azienda Ospedaliera Sant'Anna e San Sebastiano (Other); Azienda Ospedaliera, Ospedale Civile di Legnano (Other)
Responsible Party: Principal Investigator, Marco Ferlini, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXO_01; 2018-001065-17 (EudraCT Number)
Record Dates: First submitted 2020-03-06; First posted 2020-03-11 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: ST-elevation Myocardial Infarction
Keywords: Myocardial Infarction; Percutaneous Coronary Intervention; Evolocumab; Cardiac Magnetic Resonance
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Evolocumab (Experimental): Evolocumab administration in the acute phase of ST elevation myocardial infarction
  Interventions: Biological: Evolocumab
- Standard of care (No Intervention)

INTERVENTIONS:
Biological: Evolocumab — Evolocumab 140 mg every 2 weeks plus Standard of Care, including optimal lipid lowering treatment (high dose of statin ± ezetimibe)
  Other Names: Repatha
  Arms: Evolocumab

SUMMARY:
This is a prospective, multi-centre, open label, randomised study of Phase II that enrolls patients hospitalized with a diagnosis of ST-elevation myocardial infarction (STEMI), comparing Evolocumab versus Standard of Care.

DETAILED DESCRIPTION:
Primary objective of the study is to assess whether early evolocumab administration reduces infarct size in patients with STEMI undergoing primary PCI.

At least 150 patients will be enrolled to investigate the efficacy and safety of evolocumab administration in the acute phase of STEMI.

Patients will be followed for 1 year after the enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Chest pain or equivalent lasting > 20 minutes
* ST elevation myocardial infarction scheduled for primary PCI
* Signed written informed consent

Exclusion Criteria:

* Previous myocardial infarction
* Previous percutaneous or surgical myocardial revascularization
* Ongoing treatment with any statin or ezetimibe
* History of congestive heart failure
* Cardiogenic shock at presentation
* Known Pregnancy
* Women of Childbearing Age
* Known major active infection or major hematologic, renal, hepatic, or endocrine dysfunction
* Malignancy (except non-melanoma skin cancer, cervical in situ carcinoma, breast ductal carcinoma in situ, stage 1 prostate carcinoma) within the last 10 years
* Patients with hypersensitivity to the active substance (evolocumab) or to any of its excipients
* Inability to attend the scheduled clinical evaluation and laboratory tests
* Inability to undergo the pharmacological treatment or other procedures of the study
* Currently enrolled in another investigational drug study, or < 30 days/<5 half-life since ending another investigational drug study(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Infarct Size reduces infarct size in patients with STEMI undergoing primary PCI | 6 months Visit
  • Myocardial salvage index (MSI) at 6 months evaluated with cardiac magnetic resonance (CMR)

SECONDARY OUTCOMES:
Inflammatory Cytokine Response | 6 months Visit
  Absolute changes of hs-C reactive protein, Interleukin 1, 6 and10, and alfa Tumor Necrosis Factor
Cholesterol LDL levels | 6 months Visit
  Absolute and percentage changes in c-LDL levels
Major adverse cardiovascular events | 12 months Visit
  Rate of composite cardiovascular death, MI or stroke
Euroqol 5-dimension questionnaire | 12 months Visit
  Euroqol 5-dimension questionnaire (minimum value 0, and maximum value 100)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, PV, Italy